CLINICAL TRIAL: NCT07034079
Title: The Impact of Palatal Rugae Addition to Complete Dentures on Patients' Satisfaction and Oral Health Related Quality of Life: A Randomized Crossover Clinical Trial
Brief Title: The Impact of Palatal Rugae Addition to Complete Dentures on Patients' Satisfaction and Oral Health Related Quality of Life
Acronym: Palatal rugae
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Collaborators: School of dentistry (Unknown)
Responsible Party: Principal Investigator, Chawla Rashmi, Resident, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SOD/12345
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Edentulism
Keywords: Palatal rugae; Oral health impact profile; Edentulism; complete denture
MeSH Terms: interventions — Denture, Complete

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with palatal rugae initially (Experimental): Received maxillary complete denture with palatal rugae first, followed by a smooth polished palatal surface denture after a 2-month adaptation period.
  Interventions: Device: complete dentures
- without palatal rugae initially (Experimental): Received a smooth polished palatal surface denture first, followed by a rugae-enhanced denture after a 2-month adaptation period.
  Interventions: Device: complete dentures

INTERVENTIONS:
Device: complete dentures — Participants were randomly allocated into two intervention sequences using a computer-generated randomization list. The two sequences were:
  * Group A: Received maxillary complete denture with palatal rugae first, followed by a smooth polished palatal surface denture after a 2-month adaptation period.
  * Group B: Received a smooth polished palatal surface denture first, followed by a rugae-enhanced denture after a 2-month adaptation period.

SUMMARY:
In conventional maxillary complete dentures, the palatal surface is typically smooth and polished, lacking the natural anatomy of the palatal rugae. While this design facilitates ease of cleaning, it may compromise the functional feedback required for speech and other oral functions. Since the palatal rugae contain mechanoreceptors essential for guiding the tongue during phonation and mastication, replicating these structures may enhance oral function and patient adaptation.

Given the variation in clinical outcomes reported in prior studies, a randomized crossover clinical trial is warranted to assess the impact of adding anatomically replicated palatal rugae to complete dentures.

DETAILED DESCRIPTION:
In conventional maxillary complete dentures, the palatal surface is typically smooth and polished, lacking the natural anatomy of the palatal rugae. While this design facilitates ease of cleaning, it may compromise the functional feedback required for speech and other oral functions. Since the palatal rugae contain mechanoreceptors essential for guiding the tongue during phonation and mastication, replicating these structures may enhance oral function and patient adaptation.

Given the variation in clinical outcomes reported in prior studies, a randomized crossover clinical trial is warranted to assess the impact of adding anatomically replicated palatal rugae to complete dentures. This study aims to evaluate whether incorporating palatal rugae can improve patient satisfaction and oral health-related quality of life when compared to conventional dentures with a smooth palatal surface.

By assessing patient-reported outcomes in a controlled and systematic manner, this research will contribute valuable evidence toward optimizing complete denture design for better functional and psychological outcomes in edentulous patients.

OBJECTIVE

• To compare conventional complete maxillary dentures with a smooth, polished palatal surface to those incorporating anatomical palatal rugae, in terms of patient-reported outcomes and oral health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 45-80 years.
* Completely edentulous for at least 3 months.
* Seeking new complete maxillary dentures for the first time.
* Provided written informed consent
* Motivated and compliant patients, willing to return for follow-up (helps reduce attrition bias)
* Patients with Class I maxillomandibular relationship

EXCLUSION CRITERIA

* Patients with severe systemic diseases or neuromuscular dysfunction.
* Presence of mental or auditory impairment.
* History of oral pathology, xerostomia, or ankyloglossia (tied tongue).
* Previous or experienced complete denture wearers.
* Patient with strong gag reflex

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
General satisfaction | 2 months
  VAS score comparison between palatal contours

SECONDARY OUTCOMES:
Satisfaction with eating, taste, speech, phonetics, ease of cleaning | 2 months
  OHIP

IPD SHARING:
Plan to Share IPD: Undecided